CLINICAL TRIAL: NCT01530750
Title: READ-POAF Pilot Study. The Use of the Reveal XT as Device for Postoperative Atrial Fibrillation Detection After Cardiac Surgery
Brief Title: READ-POAF Pilot Studies Postoperative Atrial Fibrillation After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL37204.060.11
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Atrial Fibrillation
Keywords: postoperative atrial fibrillation; internal loop recorder; risk factors; coronary artery bypass surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post cardiac surgery

SUMMARY:
Postoperative atrial fibrillation after coronary artery bypass grafting will be monitored up to 1 year after the procedure by implanting a Reveal XT internal loop recorder two weeks before the surgery. Frequency, burden, and possible risk factors will be described.

During the operation direct contact epicardial mapping will be performed and tissue samples will be collected to identify an electrophysiological and a structural substrate for development of AF.

DETAILED DESCRIPTION:
Background of the study:

Postoperative atrial fibrillation (POAF) after cardiac surgery is a common (1 in 4) complication and associated with morbidity and mortality. Not all episodes of AF are noticed and detected, especially after discharge. several studies have shown high mortality in POAF patients, suggesting a progression in AF frequency.

Objective of the study:

To investigate the real incidence and burden of POAF. Afterwards a risk stratification of POAF is made. To identify a structural and electrophysiological substrate for the development of POAF and new onset AF during follow up.

Study design:

140 patients will receive a Reveal device. After 3 and 12 months data will be subtracted from the device. 100 of these patient will undergo additional mapping and tissue biopsies during operation.

Study population:

All patients undergoing cardiac surgery without a history of AF and without a pacemaker will be invited to participate in the study.

Primary study parameters/outcome of the study:

Incidence of POAF until 3 months after CABG.

Secondary study parameters/outcome of the study:

Incidence of POAF until 12 months after CABG. Determine risk factors for early and late POAF. Detect pre-operative (unnoticed) episodes of AF.

Determine a substrate for development of AF.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

There is a small risk of minor complications (hemorrhage and infection of the pocket).The device can be explanted easily if necessary. Ther is a burden of the im- and explantation of the device (local anesthesia, approx. 20 minutes). Patient will have to visit the out-hospital clinic twice.

The operation will be prolonged by 30 minutes due to mapping.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing non emergency surgery
* Sinus rhythm on initial visit

Exclusion Criteria:

* History of atrial fibrillation
* Internal pacemaker

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: those patients undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation (AF) | 3 months
  frequency, frequency distribution, and burden of AF

SECONDARY OUTCOMES:
atrial fibrillation (AF) | 12 months
  frequency, frequency distribution, burden of AF, AF substrate

CONTACTS AND LOCATIONS:
Overall Officials: Bart van Straten, MD, PhD, Principal Investigator — CZE; Sander Bramer, MD, Study Director — CZE; Jos Maessen, MD. PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - Maastricht University Medical Center, Maastricht

REFERENCES:
- [Derived] Bidar E, Zeemering S, Gilbers M, Isaacs A, Verheule S, Zink MD, Maesen B, Bramer S, Kawczynski M, Van Gelder IC, Crijns HJGM, Maessen JG, Schotten U. Clinical and electrophysiological predictors of device-detected new-onset atrial fibrillation during 3 years after cardiac surgery. Europace. 2021 Dec 7;23(12):1922-1930. doi: 10.1093/europace/euab136. PMID 34198338